CLINICAL TRIAL: NCT06194175
Title: Evolution of Alcohol Consumption Patterns After Bariatric Surgery and Associated Factors
Brief Title: Alcohol Consumption After Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Esin ER, Principal Investigator, University of Liege
Other Study IDs: 2023-043 (CHU de Liège)
Record Dates: First submitted 2023-12-02; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Bariatric Surgery; Obesity; Alcohol Drinking
Keywords: bariatric surgery; obesity; alcohol; predictor; longitudinal
MeSH Terms: conditions — Obesity; Alcohol Drinking | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing bariatric surgery: 350 adults (1) suffering from obesity, with a body mass index (BMI) greater than or equal to 40, or a BMI greater than or equal to 35 with at least one obesity-related comorbidity; (2) and whose candidacy for bariatric surgery has been accepted (i.e. who have obtained an operation date).
  Participants are recruited from four hospitals practicing bariatric surgery in Belgium.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Participants whose application for bariatric surgery was accepted, regardless of the type of surgical intervention (e.g., sleeve gastrectomy, Roux-en-Y Gastric Bypass).
  This longitudinal study includes five measurement times: before surgery and then, 6 months, one year, one and a half years and two years after surgery. At each measurement time, participants are asked to respond to a set of online questionnaires. Responses are anonymous.

SUMMARY:
A large body of studies indicate an increase in alcohol use disorder (AUD) rates after bariatric surgery. However, little information exists on the evolution of other drinking patterns after surgery and the psychological predictors of problematic drinking postoperatively. The identification of these factors is necessary for the implementation of prevention strategies regarding postoperative problematic alcohol use. The aim of this research is to examine the evolution of various drinking patterns after bariatric surgery as well as the psychological factors associated with AUD and an increase in postoperative alcohol consumption.

DETAILED DESCRIPTION:
Obesity affects 15.9% of the Belgian population and remains a difficult disease to treat with traditional weight loss interventions. Its high prevalence and the negative consequences it entails make it a public health concern. Bariatric surgery is associated with long-term weight loss and an improvement in obesity-related comorbidities. However, despite its success in achieving significant and lasting weight loss, numerous studies raise the emergence of unpleasant psychosocial problems after the operation, including an increase of regular alcohol consumption and prevalence of AUD. Some of these studies are longitudinal and include large samples. For example, in a prospective multicenter study, King et al., (2017) found that more than 20% of patients with a bariatric surgery present symptoms of AUD within five years after surgery. Moreover, some studies suggest that, among patients with postoperative AUD, some had never suffered from alcohol problems before surgery.

Given the severe negative consequences of AUD for the individuals who suffer from it, their family and the society, better understanding the factors involved in postoperative alcohol use problems is necessary. However, little is known about predictors of post-bariatric surgery AUD. Known risk factors are: male gender, smoking, regular alcohol consumption before surgery, younger age, recreational drug use, lower sense of belonging and ADHD symptoms. Information is lacking about the psychological risk factors for postoperative AUD and regarding the evolution of problematic drinking patterns other than AUD after surgery.

Given the previously cited gaps in the scientific literature, the present research's aims are to study the evolution of different drinking patterns after bariatric surgery as well as the psychological factors associated with AUD and increased alcohol consumption postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older at the time of surgery
* Having a body mass index (BMI) greater than or equal to 40 or a BMI greater than or equal to 35 with at least one obesity-related comorbidity
* Having a scheduled surgery date
* Fluency in French speaking
* Being able to complete the questionnaires, i.e. have access to a computer or a smartphone

Exclusion Criteria:

* Being a minor at the time of the operation
* Having difficulty reading or understanding French.
* Not having access to a computer or a smartphone to answer the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (1) suffering from obesity, with a body mass index (BMI) greater than or equal to 40, or a BMI greater than or equal to 35 with at least one obesity-related comorbidity; (2) and whose candidacy for bariatric surgery has been accepted (i.e. who have obtained an operation date).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption and alcohol use disorder | Before bariatric surgery and 6 months, one year, one and a half years and two years after surgery.
  Alcohol consumption and presence of alcohol use disorder assessed using the Alcohol Use Disorders Identification Test (AUDIT). Scores on the AUDIT range from 0 to 40, with higher scores indicating more problematic alcohol use.
Binge drinking | Before bariatric surgery and 6 months, one year, one and a half years and two years after surgery.
  Frequency of binge drinking as evaluated by a three item questionnaire.
Alcohol Intoxication | Before bariatric surgery and 6 months, one year, one and a half years and two years after surgery.
  Frequency of alcohol intoxication assessed by a single item.
Antecedents of alcohol use problems | Before surgery only.
  Assessment of the lifetime presence of alcohol problems using the CAGE questionnaire (CAGE as an acronym for "Cut down drinking", "Annoyed by criticism", "Guilty feelings" and "Eye-opener").This questionnaire is made up of 4 items to which participants can respond on a binary scale ("yes" or "no"). Two or more "yes" answers indicate an alcohol abuse problem.
Drinking Motives | Before bariatric surgery and 6 months, one year, one and a half years and two years after surgery.
  Assessment of reasons for consuming alcohol using the Drinking Motives Questionnaire - Revised Short Form. This questionnaire is composed of 12 items and 4 subscales assessing four types of motivation to drink. Scores on each of the subscales range from 3 to 9, with higher scores indicating more motivations to drink.
Sensitivity to alcohol | At 6 months and one year after surgery.
  Single-question assessment of the extent to which participants perceive a change in their response to alcohol following bariatric surgery.

SECONDARY OUTCOMES:
Binge eating | Before bariatric surgery and one and two years post-surgery.
  Assessment of binge eating behaviors using the Binge Eating Scale. Scores on this scale range from 0 to 46, with a higher score indicating a higher levels of binge eating. A score greater than or equal to 18 on this scale indicates binge eating disorder.
Emotional eating | Before bariatric surgery and one and two years post-surgery.
  Assessment of emotional eating through the "emotional eating" subscale of the Dutch Eating Behavior Questionnaire. Scores on this subscale range from 13 to 65, with higher scores indicating a greater tendency toward emotional eating.
Grazing | Before bariatric surgery and one and two years post-surgery.
  Assessment of grazing behaviors through a single question.
Emotion regulation | Before bariatric surgery and one and two years post-surgery.
  Assessment of emotional regulation using the Difficulties in Emotion Regulation Scale. It includes 6 subscales (i.e., nonacceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies and lack of emotional clarity). A total score is calculated as well as scores for each subscale. Higher scores suggest higher levels of emotional regulation deficits.
Experiential Avoidance | Before bariatric surgery and one and two years post-surgery.
  Assessment of experiential avoidance using the Brief Experiential Avoidance Questionnaire. Scores on this scale range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
Impulsivity | Before bariatric surgery and one year post-surgery.
  Assessment of impulsivity through a short version of the UPPS-P Impulsive Behavior Scale. This scale includes 5 subscales: negative urgency, positive urgency, lack of premeditation, lack of perseverance, and sensation seeking. Higher scores on these subscales indicate higher levels of impulsivity.
Anxiety | Before bariatric surgery and 6 months, one year, one and a half years and two years after surgery.
  Assessment of anxiety using the "Anxiety" subscale of the Hospital Anxiety and Depression Scale.This subscale has 7 items. Scores vary between 0 and 21. A score greater than or equal to 8 is an indicator of anxiety.
Depression | Before bariatric surgery and 6 months, one year, one and a half years and two years after surgery.
  Assessment of depressive symptoms using the "Depression" subscale of the Hospital Anxiety and Depression Scale.This subscale has 7 items. Scores vary between 0 and 21. A score greater than or equal to 8 is an indicator of depressive symptoms.

OTHER OUTCOMES:
Sociodemographic data | These questions are only asked at baseline, before bariatric surgery. They will be used to provide the description of the participant's characteristics and to control their effects while conducting some statistical analyses.
  Questions relating to age, gender, professional, marital status, etc.
Type of surgery | Before surgery only.
  One question regarding the type of surgical procedure the patient will undergo.
Weight | Before bariatric surgery and 6 months, one year, one and a half years and two years after surgery.
  Weight in kilograms.
Height | Before surgery only.
  Height in meters.

CONTACTS AND LOCATIONS:
Overall Officials: ER Esin, Principal Investigator — University of Liège (Research Unit for a life-Course perspective on Health & Education)
Locations (4):
- Belgium (4):
  - Centre Hospitalier Interrégional Edith Cavell - site Delta, Auderghem
  - Grand Hôpital de Charleroi, Charleroi
  - Centre Hospitalier Universitaire de Liège, Liège
  - Centre Hospitalier Universitaire CHU UCL Namur - site Sainte-Elisabeth, Namur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arterburn DE, Telem DA, Kushner RF, Courcoulas AP. Benefits and Risks of Bariatric Surgery in Adults: A Review. JAMA. 2020 Sep 1;324(9):879-887. doi: 10.1001/jama.2020.12567. PMID 32870301
- [Background] Cuellar-Barboza AB, Frye MA, Grothe K, Prieto ML, Schneekloth TD, Loukianova LL, Hall-Flavin DK, Clark MM, Karpyak VM, Miller JD, Abulseoud OA. Change in consumption patterns for treatment-seeking patients with alcohol use disorder post-bariatric surgery. J Psychosom Res. 2015 Mar;78(3):199-204. doi: 10.1016/j.jpsychores.2014.06.019. Epub 2014 Sep 7. PMID 25258356
- [Background] Ibrahim N, Alameddine M, Brennan J, Sessine M, Holliday C, Ghaferi AA. New onset alcohol use disorder following bariatric surgery. Surg Endosc. 2019 Aug;33(8):2521-2530. doi: 10.1007/s00464-018-6545-x. Epub 2018 Oct 22. PMID 30350107
- [Background] Ivezaj V, Benoit SC, Davis J, Engel S, Lloret-Linares C, Mitchell JE, Pepino MY, Rogers AM, Steffen K, Sogg S. Changes in Alcohol Use after Metabolic and Bariatric Surgery: Predictors and Mechanisms. Curr Psychiatry Rep. 2019 Aug 13;21(9):85. doi: 10.1007/s11920-019-1070-8. PMID 31410716
- [Background] King WC, Chen JY, Courcoulas AP, Dakin GF, Engel SG, Flum DR, Hinojosa MW, Kalarchian MA, Mattar SG, Mitchell JE, Pomp A, Pories WJ, Steffen KJ, White GE, Wolfe BM, Yanovski SZ. Alcohol and other substance use after bariatric surgery: prospective evidence from a U.S. multicenter cohort study. Surg Obes Relat Dis. 2017 Aug;13(8):1392-1402. doi: 10.1016/j.soard.2017.03.021. Epub 2017 Mar 31. PMID 28528115
- [Background] King WC, Chen JY, Mitchell JE, Kalarchian MA, Steffen KJ, Engel SG, Courcoulas AP, Pories WJ, Yanovski SZ. Prevalence of alcohol use disorders before and after bariatric surgery. JAMA. 2012 Jun 20;307(23):2516-25. doi: 10.1001/jama.2012.6147. PMID 22710289
- [Background] sciensano.be [Online]. Numbers ; [cited 2 déc 2023]. Available : https://www.sciensano.be/en/health-topics/obesity/numbers
- [Background] Spadola CE, Wagner EF, Dillon FR, Trepka MJ, De La Cruz-Munoz N, Messiah SE. Alcohol and Drug Use Among Postoperative Bariatric Patients: A Systematic Review of the Emerging Research and Its Implications. Alcohol Clin Exp Res. 2015 Sep;39(9):1582-601. doi: 10.1111/acer.12805. Epub 2015 Aug 4. PMID 26241357
- [Background] Wiedemann AA, Saules KK, Ivezaj V. Emergence of New Onset substance use disorders among post-weight loss surgery patients. Clin Obes. 2013 Dec;3(6):194-201. doi: 10.1111/cob.12034. Epub 2013 Oct 15. PMID 25586736